CLINICAL TRIAL: NCT06198985
Title: The Effect of Dynamic Balance Exercises Added to Current Medical Treatment on Balance in Patients With Ankylosing Spondylitis.
Brief Title: The Effect of Dynamic Balance Exercises on Balance in Patients With Ankylosing Spondylitis.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hakan Alkan (Other)
Responsible Party: Sponsor-Investigator, Hakan Alkan, Clinical Professor, Pamukkale University
Organization: Pamukkale University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PamukkaleU-Karaköseli-002
Record Dates: First submitted 2023-12-27; First posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-12

CONDITIONS: Ankylosing Spondylitis
Keywords: Tecnobody; Ankylosing spondylitis; Balance
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dynamic balance exercise with tecnobody prokin 252 balance device added to current medical treatment (Experimental): Dynamic balance exercises: The treatment will be performed in 3 days a week for 6 weeks. Each exercise will last 30 minutes. It will take 18 sessions in total. These exercises include 14 balance exercise movements performed on tecnobody prokin 252 balance device.
  Interventions: Procedure: Dynamic balance exercise with tecnobody prokin 252 balance device
- Group receiving current medical treatment (No Intervention): Participants in this group will receive only current medical treatment.

INTERVENTIONS:
Procedure: Dynamic balance exercise with tecnobody prokin 252 balance device — Dynamic balance exercise with tecnobody prokin 252 balance device
  Arms: Dynamic balance exercise with tecnobody prokin 252 balance device added to current medical treatment

SUMMARY:
The aim of the study is to investigate the effect of dynamic balance exercises added to current medical treatment on balance in patients with ankylosing spondylitis.

DETAILED DESCRIPTION:
The study was planned as a randomized controlled study. Forty participants with a clinically confirmed diagnosis of AS according to ASAS criteria will be recruited from the PAU Department of Physical Medicine and Rehabilitation (PMR). These participants who meet the inclusion and exclusion criteria will be randomly divided into 2 groups.

The trial will be carried out at Pamukkale University Department of Physical Medicine and Rehabilitation between January 2024 and July 2025. The local ethics committee approved the study. All participants will be informed about the purpose and content of the study and will sign written consent to participate in the study.

Participant's age, gender, body mass index, education, occupation, medications, duration of diagnosis, comorbidity, functional status and pain will be questioned and recorded.

Group1: Group receiving dynamic balance exercise with tecnobody prokin 252 balance device added to current medical treatment (Intervention group) The first group will be given dynamic balance exercises with the tecnobody prokin 252 device and participants will continue their current medical treatment. These dynamic balance exercises will be performed in 3 days a week for 6 weeks. Each exercise will last 30 minutes. It will take 18 sessions in total. These exercises include 14 balance exercise movements performed on tecnobody prokin 252 balance device (manufactured in Italy).

Group 2: Group receiving current medical treatment (control group) Participants in this group will receive only current medical treatment. Care will be taken not to change the medical treatments of the participants during the study.

All participants will be evaluated with the following evaluation parameters before the treatment and at the end of 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18 to 65 years with a clinical diagnosis of ankylosing spondylitis according to ASAS criteria
* To have the ability to give written informed consent
* Having the ability to understand procedures

Exclusion Criteria:

* Visual and vestibular system diseases that may affect balance
* Neurological or orthopedic diseases that may affect balance (Parkinson's disease, history of stroke, presence of knee or hip prosthesis, previous fracture sequelae, foot problems, etc.)
* Individuals with severe mental and sensory problems
* History of balance exercise and/or spine surgery in the last 6 months
* Pregnancy or breastfeeding
* Over 150 kg

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Dynamic balance measurements | a day before rehabilitation
  The TecnoBody Prokin 252 system was used to assess balance in the standing position for all participants. This equipment provides data on average track error and stability index.
Dynamic balance measurements | 6 weeks after the start of rehabilitation
  The TecnoBody Prokin 252 system was used to assess balance in the standing position for all participants. This equipment provides data on average track error and stability index.

SECONDARY OUTCOMES:
ASQoL | a day before rehabilitation
  A disease-specific, patient-completed outcome measure for patients with AS. The scale consists of 18 questions with two answers as 0 'no' and 1 'yes' for each item. The total score ranges from 0-18, with a high score indicating good quality of life.
ASQoL | 6 weeks after the start of rehabilitation
  A disease-specific, patient-completed outcome measure for patients with AS. The scale consists of 18 questions with two answers as 0 'no' and 1 'yes' for each item. The total score ranges from 0-18, with a high score indicating good quality of life.
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | a day before rehabilitation
  It consists of 6 VAS measures of fatigue, spinal and peripheral joint pain, tenderness and morning stiffness. Morning stiffness is measured in terms of both severity and duration. The mean score for the two questions on morning stiffness is calculated and summed with the scores for the other questions. The BASDAI score is obtained by converting the total value into a 0-10 scale. Below four is considered inactive disease and four and above is considered active disease.
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | 6 weeks after the start of rehabilitation
  It consists of 6 VAS measures of fatigue, spinal and peripheral joint pain, tenderness and morning stiffness. Morning stiffness is measured in terms of both severity and duration. The mean score for the two questions on morning stiffness is calculated and summed with the scores for the other questions. The BASDAI score is obtained by converting the total value into a 0-10 scale. Below four is considered inactive disease and four and above is considered active disease.
Bath Ankylosing Spondylitis Functional Index (BASFI) | a day before rehabilitation
  It is a quick, easy-to-administer functional index consisting of ten items developed to assess the functional status of patients. The total BASFI score is evaluated between 0-10.
Bath Ankylosing Spondylitis Functional Index (BASFI) | 6 weeks after the start of rehabilitation
  It is a quick, easy-to-administer functional index consisting of ten items developed to assess the functional status of patients. The total BASFI score is evaluated between 0-10.
Bath Ankylosing Spondylitis Metrology Index (BASMI) | a day before rehabilitation
  It is used to measure the level of spinal mobility of patients. The higher the BASMI score, the more severe the patient's limitation of movement.
Bath Ankylosing Spondylitis Metrology Index (BASMI) | 6 weeks after the start of rehabilitation
  It is used to measure the level of spinal mobility of patients. The higher the BASMI score, the more severe the patient's limitation of movement.

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Alkan, Study Director — Pamukkale University

IPD SHARING:
Plan to Share IPD: No